CLINICAL TRIAL: NCT03081780
Title: Open Label Dose Escalation Trial of an Adaptive Natural Killer (NK) Cell Infusion (FATE-NK100) With Subcutaneous IL-2 in Adults With Refractory or Relapsed Acute Myelogenous Leukemia (AML)
Brief Title: Open Label NK Cell Infusion (FATE-NK100) With Subq IL-2 in Adults With AML
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016LS153
Record Dates: First submitted 2017-03-06; First posted 2017-03-16 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Refractory Acute Myelogenous Leukemia; Relapsed Acute Myelogenous Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FATE NK-100 (Experimental)
  Interventions: Biological: FATE-NK100

INTERVENTIONS:
Biological: FATE-NK100 — Preparative regimen:
  * Fludarabine 25 mg/m2 x 5 days start Day -6
  * Cyclophosphamide 60 mg/kg x 2 days on Day -5 and -4
  Apheresis cell collection (collected from the Donor Day - 8) will be enriched for FATE-NK100 per CMC. IL-2 at 6 million IU subcutaneously (SC) every other day (EOD) for 6 doses with Dose 1 on Day 0 (no sooner than 4 hours post NK cells) and last dose no later than Day +12.

SUMMARY:
This is a Phase I open-label dose escalation study of a single infusion of FATE-NK100 and a short course of subcutaneous interleukin-2 (IL-2) administered after lymphodepleting chemotherapy (CY/FLU) in subjects with refractory or relapsed acute myelogenous leukemia (AML). FATE-NK100 is a natural killer (NK) cell product that is enriched for NK cells with an "adaptive", or human cytomegalovirus (CMV)-induced, phenotype. The NK cell product is comprised of peripheral blood (PB) leukocytes sourced from a related donor (HLA-haploidentical or better but not fully HLA-matched) that is seropositive for cytomegalovirus (CMV+), and enriched for adaptive NK cells by depletion of CD3+ (T-lymphocytes) and CD19+ (B-lymphocytes) cells followed by ex-vivo culture expansion.

ELIGIBILITY:
Inclusion Criteria:

- ≥18 but ≤ 70 years of age

* Diagnosis of acute myeloid leukemia (AML) and meets one of the following disease criteria:

  * Primary induction failure:

  ** De Novo AML: no CR after 2, 3 or 4 induction attempts with high dose chemotherapy
  * Secondary AML (from MDS or treatment related): no CR after 1, 2 or 3 cycles of high dose chemotherapy

    * Relapsed:
  * Not in CR after 1 or 2 cycles of standard re-induction therapy
  * Relapse diagnosed at the time of the 6 months post-HCT standard of care follow-up or later (i.e. based on bone marrow biopsy performed Day +170 or later) and without evidence of graft versus host disease (GVHD)

    * For patients > 60 years of age, the minimum of 1 cycle of standard chemotherapy is not required.
* Available HLA-matched or better but not fully HLA-matched (2/4 or 3/4 antigens) related donor (aged 18 to 75 years) with donor/recipient match based on a minimum of intermediate resolution DNA based Class I typing of the A and B locus who is CMV seropositive.
* Karnofsky Performance Status ≥ 60%
* Adequate organ function within 14 days of study registration (28 days for pulmonary and cardiac) defined as:

  * Creatinine: Estimated glomerular filtration rate (eGFR) ≥ 50 mL/min/1.73m^2 per current institutional calculation formula
  * Hepatic: AST and ALT ≤ 3 x upper limit of institutional normal
  * Pulmonary Function: oxygen saturation ≥ 90% on room air; PFT's required only if symptomatic or prior known impairment - must have pulmonary function >50% corrected DLCO and FEV1
  * Cardiac Function: LVEF ≥ 40% by echocardiography or MUGA
  * No symptomatic active conduction system abnormalities
* Able to be off prednisone or other immunosuppressive medications for at least 3 days prior to FATE-NK100 cell infusion (excluding preparative regimen premedications)
* Sexually active females of child bearing potential and males with partners of child bearing potential must agree to use effective contraception during therapy and for 4 months after completion of therapy
* Voluntary written consent prior to the performance of any research related procedures

Arm Specific Inclusion Criteria

High-Risk aGVHD (ARM 1):

- Pediatric or adult (ages 0-76 years) HCT recipients with high-risk acute GVHD, as determined either by the refined MN acute GVHD risk score [28]: http://z.umn.edu/MNAcuteGVHDRiskScore OR high risk on the basis of blood biomarkers (Ann Arbor Score 3) [31]. Patients in this arm must start treatment within the first 7 days after onset of high-risk aGVHD.

or

Steroid- Dependent aGVHD (ARM 2A):

- Pediatric or adult (ages 0-76 years) HCT recipient with grade II-IV steroid-dependent acute GVHD, defined as any one of the following: Flare of acute GVHD of at least grade II/IV severity within 8 weeks of tapering down or (off of) immunosuppression for acute GVHD, with the flare occurring on ≤0.5 mg/kg prednisone. This can include late-onset aGVHD and overlap syndrome.

or

Steroid-Refractory aGVHD (ARM 2B):

- Pediatric or adult (ages 0-76 years) HCT recipient with grade II-IV steroid refractory acute GVHD, defined as any one of the following:

* No response of acute GVHD after at least 4 days of systemic corticosteroids of at least 2 mg/kg prednisone or equivalent
* Progression of acute GVHD within 3 days of systemic corticosteroids of at least 2 mg/kg prednisone or equivalent
* Failure to improve to at least grade II acute GVHD after 14 days of systemic corticosteroids, with initial doses of at least 2 mg/kg prednisone or equivalent
* Flare of acute GVHD of at least grade II/IV severity while on steroids at a dose >0.5/mg/kg/day. This can include late-onset aGVHD and overlap syndrome.

Exclusion Criteria:

* Myocardial Infraction (MI) within the previous 6 months
* Acute leukemias of ambiguous lineage
* Pregnant or breastfeeding - The agents used in this study include those that fall under Pregnancy Category D - have known teratogenic potential. Women of child bearing potential must have a negative pregnancy test at screening
* History of or known active CNS involvement with AML
* Active autoimmune disease requiring systemic immunosuppressive therapy
* History of severe asthma and currently on chronic systemic medications (mild asthma requiring inhaled steroids only is eligible)
* New or progressive pulmonary infiltrates on screening chest X-ray or chest CT scan unless cleared for study by Pulmonary. Infiltrates attributed to infection must be stable/improving (with associated clinical improvement) after 1 week of appropriate therapy (4 weeks for presumed or documented fungal infections).
* Uncontrolled bacterial, fungal or viral infections including HIV-1/2 or active hepatitis C/B - chronic asymptomatic viral hepatitis is allowed
* Received any investigational agent within the 14 days before the start of study treatment (1st dose of fludarabine)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 3 months
  Maximum FATE-NK100 dose which could be given to 3 participants such that not more than 1 participant experienced a DLT.

SECONDARY OUTCOMES:
Clinical activity by CR/CRp leukemia clearance | Day +42
  Incidence of CRp defined as leukemia clearance (≤5%marrow blasts and no circulating peripheral blasts)
Clinical activity by CR/CRp neutrophil recovery | Day +42
  Incidence of CRp defined as neutrophil recovery (ANC >500 cells/microliter) but with incomplete platelet recovery
In vivo expansion of NK cells | Day +14
  Incidence of in vivo expansion (≥ 100 donor derived NK cells per uL blood) of NK cells
Treatment Related Mortality (TRM) | 6 months
  Incidence of treatment related mortality (TRM)
Minimal residual disease (MRD) by bone marrow morphology | up to Day 28
  Incidence of minimal residual disease (MRD) clearance by bone marrow morphology after NK Cell infusion
Minimal residual disease (MRD) by flow cytometry | up to Day 28
  Incidence of minimal residual disease (MRD) clearance by flow cytometry after NK Cell infusion
Leukemia free survival (LFS) | 1 year
  Incidence of Leukemia free survival (LFS)
Overall survival (OS) | 1 year
  Incidence of overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Murali Janakiram, MD, MS, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Masonic Cancer Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided